CLINICAL TRIAL: NCT01837498
Title: Reversal of Neuromuscular Blockade in Thoracic Surgical Patients
Status: Completed | Type: Observational
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Glenn Murphy, Director, Clinical Research, Endeavor Health
Other Study IDs: EH13-031
Record Dates: First submitted 2013-04-17; First posted 2013-04-23 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Residual Neuromuscular Blockade
Keywords: residual neuromuscular blockade, sugammadex, neostigmine, thoracic surgery
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Neostigmine; Sugammadex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Neostigmine group: At the conclusion of the surgical procedure, neuromuscular block will be reversed with neostigmine
  Interventions: Drug: Neostigmine
- Sugammadex group: At the conclusion of the surgical procedure, neuromuscular block will be reversed with sugammadex
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Neostigmine — At the conclusion of the surgical procedure, neuromuscular block will be reversed with neostigmine
  Groups: Neostigmine group
Drug: Sugammadex — At the conclusion of the surgical procedure, neuromuscular block will be reversed with sugammadex
  Groups: Sugammadex group

SUMMARY:
The majority of patients undergoing surgery receive neuromuscular blocking agents (NMBAs) in the operating room. Reversal of neuromuscular blockade at the conclusion of a general anesthetic is accomplished with cholinesterase inhibitors (primarily neostigmine). Although these drugs are often effective in enhancing recovery of muscle strength, the onset of effect is often slow (usually 15-30 minutes). More effective neuromuscular reversal agents are needed in clinical practice to enhance surgical and anesthetic management of perioperative patients. A new reversal agent (sugammadex) will likely be approved for clinical use in the United States next year. Unlike neostigmine, sugammadex is effective in providing rapid antagonism of all levels of neuromuscular blockade (typically within 2-4 minutes). The aim of this prospective observational study is to study neuromuscular and clinical recovery in 100 consecutive thoracic surgical patients receiving neostigmine, followed by a 100 consecutive thoracic surgical patients administered sugammadex (after the drug is approved by the FDA). In addition, after data on 100 patients reversed with neostigmine is collected, the data will be analyzed to compare patients with residual block (train-of four < 0.9) and without residual block (TOF </= 0.9)

DETAILED DESCRIPTION:
Patients undergoing thoracic surgical procedures receive a general anesthetic in the operating room. As part of this general anesthetic, patients are administered a neuromuscular blocking agent (NMBA or muscle relaxant). NMBAs are used to facilitate placement of endotracheal tubes (breathing tubes), provide muscle relaxation during surgery, and prevent patient movement. Most thoracic surgeons request deep levels of muscle relaxation during operative procedures. In particular, deeper levels of neuromuscular blockade are required to prevent movement of the diaphragm (diaphragmatic contractions can interfere with the surgical procedure).

Muscle contraction occurs when the neurotransmitter acetylcholine binds to the postjunctional nicotinic acetylcholine receptor (nAChR). Non-depolarizing NMBAs inhibit neuromuscular transmission primarily by competitively antagonizing or blocking the effect of acetylcholine at the postjunctional nAChR. When high enough concentrations of NMBAs are present, binding to the nAChR occurs, thus preventing acetylcholine from activating the receptor. Binding of NMBAs to the nAChR occurs in a competitive fashion. If higher concentrations of acetylcholine are present at the neuromuscular junction, acetylcholine will attach to the postsynaptic receptor and facilitate neuromuscular transmission and muscle contraction. Conversely, if higher concentrations of nondepolarizing NMBAs are present at the neuromuscular junction, binding to the nAChR will preferentially occur, preventing muscle depolarization from occurring.

The effects of NMBAs must be reversed at the end of surgery. One mechanism of antagonizing the effects of NMBAs is to increase the concentration of acetylcholine at the neuromuscular junction. This can be accomplished using an anticholinesterase drug which inhibits the enzyme which breaks down acetylcholine at the neuromuscular junction (acetylcholinesterase). The anticholinesterase drug which is most commonly used to reverse neuromuscular blockade is neostigmine. At NorthShore University HealthSystem, all patients receiving a NMBA are reversed with neostigmine at the conclusion of the surgical procedure. There are two important limitations of anticholinesterase reversal agents, which are related to their mechanism of action as described above. First, onset of action is slow. In the presence of mild degrees of muscle relaxation (four responses to train-of-four (TOF) nerve stimulation with a peripheral nerve stimulator, also known as a TOF count of 4), adequate reversal of NMBAs takes approximately 10-15 minutes. However, in the presence of deeper neuromuscular block (one response to TOF nerve stimulation, or TOF count of 1), complete reversal takes on average 30-60 minutes. Second, profound neuromuscular blockade cannot be antagonized. If no evidence of neuromuscular recovery is present at the end of surgery (no response to peripheral nerve stimulation or a TOF count of 0), reversal agents are ineffective. In this situation, the concentration of the NMBA at the neuromuscular junction is too high (NMBA will preferentially bind to the nAChR over acetylcholine, and inhibition of acetylcholinesterase cannot raise levels of acetylcholine enough to competitively antagonize the NMBA).

Despite the routine reversal of muscle relaxants in the operating room, patients often arrive in the post anesthesia care unit (PACU) with evidence of residual muscle weakness (termed residual neuromuscular blockade). Traditionally, residual neuromuscular blockade has been measured and defined using quantitative neuromuscular monitoring devices. These devices use electrical energy to stimulate the ulnar nerve; four stimuli are provided, and the response to nerve stimulation at the thumb measured. The ratio of the fourth contraction is compared to the first contraction to generate a TOF ratio (from 0-1.0 or 0-100%). Recent data suggests that TOF ratios must recover to > 0.9 to exclude clinically significant residual neuromuscular blockade. A number of clinical studies have demonstrated that approximately 40% of patients given NMBAs in the operating room have objective evidence of muscle weakness (a TOF ratio < 0.9) on admission to the PACU. It is likely that the incidence of residual neuromuscular blockade is higher in thoracic surgical patients, since deeper levels of neuromuscular blockade are required. However, no previous studies have specifically investigated this patient population.

The presence of residual muscle weakness at the end of surgery, following tracheal extubation (removal of the breathing tube), has been associated with a number of adverse postoperative events. Patients with TOF ratios < 0.9 on admission to the PACU are at higher risk for potentially life threatening airway events, including hypoxemia (low oxygen saturation), airway obstruction, and postoperative pulmonary complications. In addition, patients with TOF ratios < 0.9 often experience unpleasant symptoms of muscle weakness, such as blurry vision, difficultly speaking and swallowing, and general weakness. Patient-perceived quality of recovery from anesthesia and surgery is also significantly lower in patients admitted to the PACU with TOF ratios < 0.9. Studies have also demonstrated that patients with TOF ratios < 0.9 take significantly longer to reach discharge criteria from the PACU, and achieve actual PACU discharge.

Improved management of neuromuscular blockade in the operating can beneficially impact both the incidence of residual neuromuscular blockade, as well as complications associated with incomplete neuromuscular recovery. For example, the use of quantitative neuromuscular monitoring, by allowing a more rational titration of NMBAs intraoperatively, has been demonstrated to reduce the risk of admission to the PACU with a TOF ratio < 0.9. Furthermore, the risk of hypoxemic events, airway obstruction, and unpleasant symptoms of muscle weakness is diminished with quantitative monitoring.

Another potential method of reducing the risk of residual neuromuscular blockade, and the complications associated with residual blockade, is through the use of a new class of NMBA reversal agent. Sugammadex is a recently developed antagonist of steroidal NMBAs that acts via a different mechanism than the anticholinesterase agents. Sugammadex (Org 25969) is a modified γ-cyclodextrin and the first selective relaxant binding agent based on an encapsulating principle for inactivation of a neuromuscular blocking agent. Sugammadex is a cylindric compound with a lipophilic cavity and a hydrophilic exterior. This structure allows the drug to take up lipophilic molecules in its core; sugammadex rapidly encapsulates steroidal NMBAs like rocuronium that are present in the circulation. Rapid encapsulation of rocuronium in the intravascular compartment results in a gradient which draws rocuronium away from the neuromuscular junction (where it is also immediately encapsulated). This principle for reversal of rocuronium- and vecuronium-induced neuromuscular block was first introduced into clinical practice in 2008 and is now available for pediatric and adult anesthesia in a majority of countries world-wide. The complex formation of sugammadex and rocuronium or vecuronium occur at all levels of neuromuscular block (profound - shallow) and displays a more rapidly-acting pharmacological profile as opposed to anticholinesterases for reversal of effect. When appropriate dosing of sugammadex is used, all levels of neuromuscular blockade can be reversed (TOF ratio > 0.9) within 2-4 minutes. Consequently, sugammadex may have the potential to markedly reduce postoperative residual neuromuscular block in the PACU. In addition, sugammadex may also reduce the incidence of adverse events related to incomplete neuromuscular recovery. Sugammadex has been extensively investigated in a large number of clinical trials and has been demonstrated to be significantly more effective and rapid in reversing all levels of neuromuscular block, when compared to neostigmine. At the present time, the safety profile of sugammadex appears similar to neostigmine, in both clinical trials and in world-wide usage (over 4 million uses, per manufacturers report).

Sugammadex may offer several potential advantages in patients undergoing thoracic surgery. Deep levels of neuromuscular blockade can be maintained until the end of the procedure, which may facilitate the performance of the surgery. Sugammadex is effective in reversing deep levels of blockade (even at a TOF count of 0 or "no twitches"), whereas neostigmine cannot antagonize deep blockade. In addition, the time in the operating room may be shortened. It is not uncommon for tracheal extubation to be delayed in this patient population due to the slow onset of effect of neostigmine when moderate levels of neuromuscular block are present at the time of reversal (TOF count of 1-3). Furthermore, patient recovery may be enhanced in the PACU if the incidence of residual block is reduced with sugammadex. The aim of this prospective observational investigation is to examine the effect of sugammadex (versus neostigmine) on recovery following thoracic surgery. In addition, after data on 100 patients reversed with neostigmine is collected, the data will be analyzed to compare patients with residual block (train-of four < 0.9) and without residual block (TOF </= 0.9) The primary outcome variable will be the incidence of residual block (measured with quantitative neuromuscular monitoring) at the time of PACU admission. Secondary outcome measures will include the incidence of residual block at tracheal extubation, the time from surgical closure until tracheal extubation, the frequency of adverse respiratory events in the PACU, the presence or absence of symptoms and signs of postoperative muscle weakness, and length of stay in the operating room and PACU.

ELIGIBILITY:
Inclusion Criteria:

* ASA I to III patients 18-80 years of age, presenting for surgery requiring maintenance of neuromuscular blockade in the operating room, will be eligible for enrollment.

Exclusion Criteria:

* Exclusion criteria include: 1) presence of an underlying neuromuscular disease 2) use of drugs known to interfere with neuromuscular transmission (antiseizure medications, anticholinesterases, magnesium sulfate) or 3) renal insufficiency (serum creatinine > 1.8 mg/dL) or renal failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients presenting for elective thoracic surgical procedures with an expected duration greater than 45 minutes will be enrolled in this study. The study is designed as a "before and after" investigation of sugammadex (data will be collected on 100 consecutive patients before sugammadex is approved by the FDA for clinical care in the United States (neostigmine used), and on 100 consecutive patients after sugammadex is approved). In addition, after data on 100 patients reversed with neostigmine is collected, the data will be analyzed to compare patients with residual block (train-of four < 0.9) and without residual block (TOF </= 0.9)
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Residual neuromuscular block (train-of-four ratio (TOF) < 0.9) | On admission to the postanesthesia care unit (PACU), up to 7 days
  The incidence of residual neuromuscular block will be calculated on arrival to the PACU

SECONDARY OUTCOMES:
Time in operating room | participants will be followed for the duration of the operating room stay, an expected average of 2 hours, up to 7 days
Hypoxemic events | participants will be followed for the duration of the PACU stay, an expected average of 2 hours, up to 7 days
  Blood oxygenation values will be measured using pulse oximetry from the time of PACU admission until discharge from the PACU
Tests of muscle weakness | 15 and 30 minutes after admission to the PACU, up to 7 days
  A standardized examination form will be used to determine the presence or absence of muscle weakness in a variety of muscle groups
Length of stay in the PACU | participants will be followed for the duration of the PACU stay, an expected average of 2 hours, up to 7 days
  The time required to meet discharge criteria and achieve actual discharge will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn S Murphy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

REFERENCES:
- [Derived] Murphy GS, Avram MJ, Greenberg SB, Bilimoria S, Benson J, Maher CE, Teister KJ, Szokol JW. Neuromuscular and Clinical Recovery in Thoracic Surgical Patients Reversed With Neostigmine or Sugammadex. Anesth Analg. 2021 Aug 1;133(2):435-444. doi: 10.1213/ANE.0000000000005294. PMID 33323787